CLINICAL TRIAL: NCT00961350
Title: A 6-Month, Phase 3, Randomized, Double-Blind, Parallel-Group, Controlled, Multi-Center Study to Evaluate the Incidence of Gastric Ulcers Following Administration of Either PA32540 or Enteric Coated Aspirin 325 mg in Subjects Who Are at Risk for Developing Aspirin-Associated Ulcers
Brief Title: A Study to Evaluate the Incidence of Gastric Ulcers Following Administration of Either PA32540 or Enteric Coated Aspirin 325 mg in Subjects Who Are at Risk for Developing Aspirin-Associated Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PA32540-301
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Ulcer
Keywords: PA32540 is proposed for the secondary prevention of cardio- and cerebrovascular events in patients at risk for developing aspirin-associated gastric ulcers.
MeSH Terms: conditions — Stomach Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PA32540 (Experimental): PA32540 tablets contain 325 mg enteric coated (EC) aspirin and 40 mg immediate-release omeprazole
  Interventions: Drug: PA32540
- EC Aspirin (Active Comparator): The comparator aspirin 325 mg enteric coated tablet (PA32540 minus omeprazole)
  Interventions: Drug: EC Aspirin 325

INTERVENTIONS:
Drug: PA32540 — PA32540 tablets contain 325 mg enteric coated (EC) aspirin and 40 mg immediate-release omeprazole
  Other Names: YOSPRALA
  Arms: PA32540
Drug: EC Aspirin 325 — The comparator aspirin 325 mg enteric coated tablet (PA32540 minus omeprazole)
  Arms: EC Aspirin

SUMMARY:
Primary: To demonstrate that PA32540 causes fewer gastric ulcers in subjects at risk for developing aspirin-associated gastric ulcers compared to enteric coated (EC) aspirin 325 mg.

ELIGIBILITY:
Inclusion criteria:

1. A. Male or non-pregnant, non-breastfeeding females who have been on daily aspirin 325 mg for at least three months and who are expected to use daily aspirin 325 mg for at least six months (Daily is defined as "at least 5 days per week"):

   AND, who are
   * 55 years of age and older; or
   * 18 - 54 years of age and have a history of a documented gastric or duodenal ulcer within the past five years.
2. A. Aspirin use should be for the secondary prevention of cardiovascular or cerebrovascular events as defined as follows:

   Have been diagnosed with or have had a history of
   * MI (myocardial infarction that has been confirmed or suspected)
   * Ischemic stroke
   * TIA (transient ischemic attack)

   Or have established, clinically significant coronary and other atherosclerotic vascular disease (meaning at high risk for surgical intervention or for MI, TIA, stroke, if left untreated), including:
   * Angina (stable or unstable)
   * Peripheral arterial disease
   * Atherosclerotic aortic disease
   * Carotid artery disease Or have had
   * CABG (coronary artery bypass graft)
   * PCI (percutaneous coronary intervention with or without stent)
   * Carotid endarterectomy
3. A. If female, subjects are eligible if they are of

   1. non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   2. childbearing potential, have a negative pregnancy test at screening, and at least one of the following applies or is agreed to by the subject:

      * Female sterilization or sterilization of male partner
      * Hormonal contraception by oral route, implant, injectable, vaginal ring
      * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year
      * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide)
      * Any other method with published data showing that the lowest expected failure rate is less than 1% per year 4. Able to understand and comply with study procedures required and able and willing to provide written informed consent prior to any study procedures being performed

Exclusion criteria:

1. Baseline endoscopy showing any gastric, esophageal or duodenal ulcer at least 3 mm in diameter with depth
2. Positive test result for H. pylori at screening 3A. Have had a revascularization procedure (i.e., Coronary Artery Bypass Graft, Percutaneous Transluminal Coronary Angioplasty, or carotid endarterectomy) less than six months prior to screening

4. Unstable hypertension as judged by the Investigator 5. Uncontrolled diabetes mellitus as judged by the Investigator 6. Unstable cardio- or cerebrovascular disease such that it would endanger the subject if they participated in the trial 7. Clinically significant valvular disease 8. Congestive heart failure or other cardiovascular symptoms according to New York Heart Association (NYHA) Functional Classification III or IV (Appendix 3) 9. History of hypersensitivity to omeprazole or to another proton pump inhibitor 10. History of allergic reaction or intolerance to aspirin and/or a history of aspirin-induced symptoms of asthma, rhinitis, and/or nasal polyps 11. History of serious UGI event, such as bleeding, perforation, or obstruction 12. Gastrointestinal disorder or surgery leading to impaired drug absorption 13. Presence of chronic or uncontrolled acute medical illness, e.g. gastrointestinal disorder (esophageal stricture, severe esophagitis, long-segment Barrett's esophagus, signs and symptoms of gastric outlet obstruction), thyroid disorder and/or infection that would endanger a subject if they were to participate in the study 14. Schizophrenia, uncontrolled bipolar disorder, or severe depression 15. History of alcoholism or drug addiction within a year prior to enrollment in the study 16. Severe hepatic dysfunction (i.e. cirrhosis or portal hypertension) 17. Blood coagulation disorder, including use of systemic anticoagulants such as warfarin or other vitamin K antagonists 18. Any condition that, in the opinion of the Investigator, may either put the subject at risk or influence the results of the study 19. Use of any excluded concomitant medication (see Section 9.2) 20. Screening laboratory ALT or AST value > two times the upper limit of normal 21A. History of renal insufficiency 22. Other than noted specifically, any screening laboratory value that is clinically significant in the Investigator's opinion and would endanger a subject if the subject was to participate in the study 23. Use of an investigational treatment in the 4 weeks before screening 24. History of malignancy, treated or untreated, within the past five years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin 25. Previous participation in another PA32540 clinical research study 26. Subjects, who are employees of the research facility, immediately related to the Principal Investigator, or are in some way under the supervision of the Principal Investigator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pozen, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PA32540: PA32540 tablets contain 325 mg enteric coated (EC) aspirin and 40 mg immediate-release omeprazole dosed once daily (QD)
- EC Aspirin: EC Aspirin 325 mg enteric coated tablet (PA32540 minus omeprazole) dosed once daily (QD)
Period: Overall Study
Arm/Group | PA32540 | EC Aspirin
Started | 265 | 265
Intent-to-Treat Population (ITT) | 265 | 265
Safety Population | 264 (1. One sub rand to PA32540 took EC-Aspirin) | 265
Completed | 218 | 198
Not Completed | 47 | 67
Not completed — Adverse Event | 18 | 33
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 3 | 3
Not completed — Misc | 16 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA32540 | EC Aspirin | Total
Number analyzed (Participants) | 265 | 265 | 530
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.2) | 65.8 (6.7) | 66.1 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 75 | 152
  Male | 188 | 190 | 378

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gastric Ulcer Confirmed by Endoscopy(EC) Aspirin 325 mg
Description: The primary efficacy endpoint was the number of subjects with gastric ulcers at any time throughout 6 months of treatment. An ulcer was defined as a mucosal break of at least 3 mm in diameter (measured by close application of open endoscopic biopsy forceps) with unequivocal crater depth. A subject is considered to have completed the study if all scheduled assessments up through the 6 month visit have been performed or if the endpoint of gastric ulcer confirmed by endoscopy has been reached.
Time Frame: 6 months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | PA32540 | EC Aspirin
Number analyzed (Participants) | 265 | 265
participants | 10 [1.8 to 6.8] | 23
Statistical Analysis 1: Comparison: PA32540 vs EC Aspirin; The primary efficacy endpoint was the proportion of subjects with gastric ulcers throughout 6 months of treatment. The primary endpoint was analyzed with the CMH test stratified by NSAID use (COX-2/Other NSAID/No) at randomization. A sample size of 250 subjects/treatment would provide 86% power to detect the difference of 8% between EC aspirin 325 mg (13%) and PA32540 (5%) with a 2-sided significance of 5%; and, provides adequate power to test the key secondary endpoints in sequential order; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel; CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization; Proportions = 3.8, 95% CI [1.8 to 6.8] — The proportion is from the PA32540 treatment group

2. Secondary Outcome: The Number of Participants With Gastric and/or Duodenal Ulcers
Description: The Number of Participants with Gastric and/or Duodenal Ulcers throughout 6 months of treatment.
Time Frame: 6 Months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | PA32540 | EC Aspirin
Number analyzed (Participants) | 265 | 265
participants | 11 | 31
Statistical Analysis 1: Comparison: PA32540 vs EC Aspirin; The cumulative proportion of subjects developing gastric ulcers and/or duodenal ulcers at 6 months was analyzed using the CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization

3. Secondary Outcome: The Number of Subjects With "Treatment Success"
Description: Those Subjects Without Gastric Ulcers and Without Upper Gastrointestinal (UGI) Adverse Events leading to discontinuation.
Time Frame: 6 Months
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | PA32540 | EC Aspirin
Number analyzed (Participants) | 265 | 265
participants | 249 | 220
Statistical Analysis 1: Comparison: PA32540 vs EC Aspirin; The cumulative proportion of subjects with Treatment Success was analyzed using the CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization

4. Secondary Outcome: The Number of Participants Discontinuing From the Study Due to NSAID-Associated Upper GI Adverse Events
Description: The Number of Participants Discontinuing from the Study Due to non-steroidal anti-inflammatory drug (NSAID)-Associated Upper GI Adverse Events during the treatment period
Time Frame: 6 months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | PA32540 | EC Aspirin
Number analyzed (Participants) | 265 | 265
participants | 6 | 22
Statistical Analysis 1: Comparison: PA32540 vs EC Aspirin; The cumulative proportion of subjects discontinuing from the study due to NSAID-associated upper GI adverse events was analyzed using the CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization

5. Secondary Outcome: The Number of Participants With Heartburn Resolution at 6 Months, ie no Heartburn Symptoms During the Last 7 Days Prior to the Visit
Description: Subjects were asked whether heartburn symptoms within the 7 days prior to the visit were:
  * none: no symptoms
  * mild: awareness of symptom, but easily tolerated
  * moderate: discomforting symptom sufficient to cause interference with normal activities (including sleep)
  * severe: incapacitating symptom, with inability to perform normal activities (including sleep) Heartburn was defined as a burning feeling rising from the stomach or lower part of the chest towards the neck.
Time Frame: 6 Months
Population: Intent to Treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | PA32540 | EC Aspirin
Number analyzed (Participants) | 265 | 265
participants | 198 | 135
Statistical Analysis 1: Comparison: PA32540 vs EC Aspirin; The proportion of subjects who had no heartburn at 6 months (regardless of the presence or absence of heartburn at baseline) was analyzed using the CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO at randomization; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; CMH test stratified by NSAID use=COX-2, other NSAID, or NSAID use=NO and by baseline heartburn severity at randomization

ADVERSE EVENTS:
Time Frame: Informed consent through 6 months plus 28 days for Serious Adverse Events and Randomization through 6 months for all non-serious adverse events.
Arm/Group | PA32540 | EC Aspirin
Serious Adverse Events (participants affected / at risk) | 16/264 | 24/265
Other Adverse Events (participants affected / at risk) | 191/264 | 224/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | PA32540 (N=264) | EC Aspirin (N=265)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0/264 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Sudden cardiac death (Cardiac disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA32540 (N=264) | EC Aspirin (N=265)
Gastritis (Gastrointestinal disorders) | 46 (51) | 44 (48)
Dyspepsia (Gastrointestinal disorders) | 35 (40) | 90 (114)
Gastritis erosive (Gastrointestinal disorders) | 27 (29) | 82 (97)
Hiatus hernia (Gastrointestinal disorders) | 27 (27) | 26 (26)
Duodenitis (Gastrointestinal disorders) | 15 (17) | 46 (47)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 8 (8)
Nausea (Gastrointestinal disorders) | 8 (8) | 7 (7)
Oesophagitis (Gastrointestinal disorders) | 8 (8) | 31 (34)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (7) | 14 (15)
Oesophageal disorder (Gastrointestinal disorders) | 7 (8) | 2 (2)
Reflux oesophagitis (Gastrointestinal disorders) | 4 (4) | 7 (7)
Erosive duodenitis (Gastrointestinal disorders) | 2 (2) | 25 (26)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 9 (9)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 10 (10)
Nasopharyngitis (Infections and infestations) | 4 (5) | 6 (6)
Bronchitis (Infections and infestations) | 3 (3) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (9)
Dizziness (Nervous system disorders) | 4 (4) | 6 (6)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that the first publication will be a multi-center publication of the study results. Following this multi-center publication, PI can publish, present or use any non-confidential study results following Sponsor review and comment.